CLINICAL TRIAL: NCT01523015
Title: Efficacy and Safety Study of the Combined Modality Therapy in Patients With Potentially Resectable, Locally Advanced Adenocarcinoma of the Esophago-gastric Junction With Preoperative Chemo- and Chemoradiation Followed by Surgical Resection
Brief Title: Efficacy and Safety Study of the Combined Modality Therapy in Adenocarcinoma of the Esophago-gastric Junction
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Lublin (Other)
Responsible Party: Principal Investigator, Tomasz Skoczylas, Principal Investigator, Medical University of Lublin
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EGC-0254/87/2011; UML-EGC-2011 (Other: UML)
Record Dates: First submitted 2012-01-25; First posted 2012-02-01 (Estimated); Last update posted 2013-02-05 (Estimated); Status verified 2013-02

CONDITIONS: Adenocarcinoma of the Gastroesophageal Junction
Keywords: Adenocarcinoma; esophago-gastric cancer; chemotherapy; chemoradiotherapy; surgery
MeSH Terms: conditions — Adenocarcinoma | interventions — Chemoradiotherapy; Docetaxel; Oxaliplatin; Fluorouracil; Radiation; Esophagectomy; Gastrectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Combined therapy (Experimental): The combined modality therapy will be consisted of preoperative chemoradiotherapy (Docetaxel, Oxaliplatin, 5-Fluorouracil, 45Gy) for type I i II cancer or preoperative chemotherapy (Docetaxel, Oxaliplatin, 5-Fluorouracil) for type III cancer and followed by surgery.
  Interventions: Other: preoperative chemo- and chemoradiotherapy
- Surgery (Active Comparator): The extent of surgery will be associated with the topographic type of carcinoma of the esophagogastric junction: type I - subtotal esophagectomy with superior gastric resection, splenectomy and two-field mediastinal lymph node dissection; type II and III - total gastrectomy with distal esophagectomy, splenectomy and D2 with mediastinal inferior lymph node dissection.
  Interventions: Procedure: Surgical resection

INTERVENTIONS:
Other: preoperative chemo- and chemoradiotherapy — 2 cycles of triple regimen chemotherapy consisting of docetaxel (75mg/m2 iv infusion), oxaliplatin (130mg/m2 iv infusion) and 5-fluorouracil (750mg/m2 iv infusion followed by fractionated irradiation (total dose 45Gy in 25 fractions of 1,8Gy) combined with chemotherapy consisting of 3 cycles of 1-day chemotherapy with docetaxel (50mg/m2 iv infusion) and oxaliplatin (85mg/m2 iv infusion
  Other Names: docetaxel,; oxaliplatin,; 5-fluorouracil,; irradiation
  Arms: Combined therapy
Procedure: Surgical resection — The extent of surgery will be associated with the topographic type of carcinoma of the esophagogastric junction: type I - subtotal esophagectomy with superior gastric resection, splenectomy and two-field mediastinal lymph node dissection; type II and III - total gastrectomy with distal esophagectomy, splenectomy and D2 with mediastinal inferior lymph node dissection.
  Other Names: esophagectomy,; gastrectomy
  Arms: Surgery

SUMMARY:
The high cancer related mortality has remained a significant issue of health care in Poland, Europe and worldwide. The decreasing incidence rate for carcinoma of the distal stomach and a marked trend of increasing incidence for adenocarcinoma of the esophago-gastric junction and esophagus has been observed in the developed countries. The most eminent drawback of majority commonly cited randomized trials is heterogenicity of cancer patient population. The epidemiological, pathological, and clinical data clearly suggest that adenocarcinoma of the esophago-gastric junction is the entirety different both from adenocarcinoma of the esophagus and adenocarcinoma of the stomach. The experience in a combined modality therapy for adenocarcinoma of the esophago-gastric junction have been extrapolated from studies on esophageal or gastric cancer, where the investigated population involved in part patients with carcinoma of the esophago-gastric junction. The proposed study has been designed to achieve the following objectives:

* The assessment of safety and efficacy of a combined modality therapy in homogenous patient population with adenocarcinoma of the esophago-gastric junction excluding individuals with adenocarcinoma of the esophagus or the stomach;
* The assessment of safety of a combined modality therapy in a form of chemo- and chemoradiotherapy related toxicity and impact of chemo- and chemoradiotherapy on postoperative morbidity or mortality rates;
* The assessment of efficacy of a combined modality therapy in a form of rate of response of the tumor to chemo- and chemoradiotherapy and a curative resection rate.
* The assessment of efficacy of a combined modality therapy in a form of cancer free survival and overall survival.

DETAILED DESCRIPTION:
Adenocarcinoma of the esophago-gastric junction (AEG) represents an aggressive disease with poor prognosis. Surgery is the traditional mainstay of treatment for patients presenting with locally advanced disease, defined as transmural invasion with or without lymph node involvement. Surgical approach may differ, but the principal is to achieve wide mural clearance, negative margins, and perform an adequate lymphadenectomy. Although surgery is the primary modality that can cure patients, the majority of patients reveal recurrence leading to death within 2 years after resection. The incidence of locoregional relapse in most series and in phase II and phase III trials ranges from 25% to 60%, and 20-30% of these patients have no evidence of distant metastases. Median survival with surgery alone for localized disease remains poor, and ranges from 13 to 19 months with 5-year survival rates at best approximately 40%. To improve a long-term outcome in patients with esophageal and gastric cancers a combined modality therapy concept has been investigating for many years. The experience in a combined modality therapy for adenocarcinoma of the esophago-gastric junction have been extrapolated from studies on esophageal or gastric cancer, where the investigated population involved in part patients with AEG.

The most eminent drawback of majority commonly cited randomized trials is heterogenicity of cancer patients population. Most of them overlap between esophageal adenocarcinoma and squamous cell carcinoma or between adenocarcinoma of the esophagus, esophagogastric junction and the stomach. When the investigators reviewed the composition of the most prominent 10 studies population including 3171 patients with easophageal and gastric cancer the investigators identified 911 (28.7%) patients with AEG. The remaining pooled population involved 1173 (36.9%) patients with adenocarcinoma of the esophagus, 598 (18.9%) patients with squamous cell carcinoma of the esophagus and 775 (24.4%) patients with adenocarcinoma of the stomach. Only 1 randomized controlled trial concerned exclusively patients with AEG. In this study preoperative chemoradiotherapy resulted in a 16% increase of 3-year survival. Although its superiority was not proven (p=0.07), these data provide evidence that preoperative chemoradiotherapy may improve survival and should be further investigated. Interestingly, the survival benefit was evident although the postoperative mortality was more than doubled (10.2% versus 3.8%) by adding chemotherapy. Although this study did not meet its accrual goals and could not provide statistical significance, the improvement in both local cancer free and overall survival suggest that preoperative chemoradiotherapy appears most valuable modality treatment to cure patients with localized AEG. As it is more than evident that major response to preoperative treatment is an important prognostic factor future trials should aim to optimize preoperative treatment by combining all treatment modalities.

All above mentioned discrepancies regarding the optimal treatment for AEG brought the investigators to an idea to design a study testing safety and efficacy of three-phase combined modality therapy accommodating induction taxane-based triple chemotherapy followed by concurrent chemoradiotherapy with 45Gy as a total dose of irradiation and subsequent surgical resection in homogenous population of patients with clearly defined AEG. Taking into account the results from recent phase II and III trials the proposed combined modality regimen suggests substantial response to the neoadjuvant therapy and promising highly effective loco-regional cancer clearance with moderate and acceptable tolerance despite a complex and extensive treatment.

ELIGIBILITY:
Inclusion Criteria:

* patients of both gender, aged more than 18, with histopathologically confirmed adenocarcinoma of the esophagogastric junction
* medically fit to undergo a major surgery with planned thoracotomy and in general condition allowing to tolerate chemo- or chemoradiotherapy (Karnofsky Performance Status ≥70, ECOG 0-1).
* Carcinoma of the esophagogastric junction defined as adenocarcinoma involving esophagogastric junction when its epicenter is localized within 5cm proximally or 5cm distally to the anatomical esophagogastric junction with subclassification to 3 topographic types (type I between 5cm and 1cm above; type II between 1cm above and 2cm below; type III between 2cm and 5cm below anatomic junction of the esophagus and the stomach).
* Potentially resectable, local or locoregional cancer with clinical staging cT2-4aN0-3M0.
* The intended number of randomized patients has been set as 100: 50 patients randomized to each therapeutic arm with assumption, that 80% of randomized patients will complete the treatment protocol.

Exclusion Criteria:

* disseminated cancer
* poor general condition (KI <70)
* adenocarcinoma of the stomach
* adenocarcinoma of the esophagus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2012-01; Primary Completion 2015-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Pathological response to treatment | 6-12 weeks after chemoradiotherapy
  Pathological response to treatment assessed as a tumor regresion grade in histopahological assessment of the surgical specimen

SECONDARY OUTCOMES:
Clinical response to treatment | 5 weeks after chemoradiotherapy
  Clinical response to treatment based on the modified RECIST criteria measured by CT
The curative resection (R0) rate | 6-12 weeks after chemoradiotherapy
  The curative resection (R0) rate defined by the assessment of proximal, distal and circumferential margins
chemoradiotherapy related toxicity | 6-12 weeks after chemoradiotherapy
  The rate and intensity of chemo- and chemoradiotherapy related toxicity
postoperative complications rate | 30 days after surgical resection
  The rate and intensity of postoperative morbidity and mortality
Overall and cancer free survival | 5 years from onset of the chemoradiotherapy
  Overall and cancer free survival
Quality of life changes | 5 years after the onset of cheemoradiotherapy
  Quality of life changes
The rate of chemo- and chemoradiotherapy dose reduction | 11 weeks during chemo- and chemoradiotherapy
  The rate of dose reduction due to chemotherapy or radiotherapy related toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Tomasz Skoczylas, MD, PhD, Principal Investigator — Second Department of General & Gastrointestinal Surgery & Surgical Oncology of the Alimentary Tract, Medical University of Lublin; Grzegorz Wallner, Professor, Principal Investigator — Second Department of General & Gastrointestinal Surgery & Surgical Oncology of the Alimentary Tract, Medical University of Lublin; Andrzej Dąbrowski, Professor, Principal Investigator — Second Department of General & Gastrointestinal Surgery & Surgical Oncology of the Alimentary Tract, Medical University of Lublin; Witold Zgodziński, MD, PhD, Principal Investigator — Second Department of General & Gastrointestinal Surgery & Surgical Oncology of the Alimentary Tract, Medical University of Lublin; Marek Majewski, MD, PhD, Principal Investigator — Second Department of General & Gastrointestinal Surgery & Surgical Oncology of the Alimentary Tract, Medical University of Lublin; Maria Mazurkiewicz, Professor, Principal Investigator — Department of Oncology, Medical University of Lublin, Lublin Oncology Center; Anna Brzozowska, MD, PhD, Principal Investigator — Department of Oncology, Medical University of Lublin, Lublin Oncology Center; Ludmiła Grzybowska-Szatkowska, MD, PhD, Principal Investigator — Department of Oncology, Medical University of Lublin, Lublin Oncology Center; Witold Krupski, Professor, Principal Investigator — Second Department of Radiology, Medical University of Lublin; Ewa Kurys-Denis, MD, PhD, Principal Investigator — Second Department of Radiology, Medical University of Lublin; Justyna Szumiło, Professor, Principal Investigator — Department of Clinical Pathomorphology, Medical University of Lublin; Agnieszka Fronczek, MD, Principal Investigator — Department of Clinical Pathomorphology, Medical University of Lublin
Locations (1):
- Second Department of General & Gastrointestinal Surgery & Oncological Surgery of the Alimantary Tract, Medical University of Lublin, Lublin, Lublin Voivodeship, Poland